CLINICAL TRIAL: NCT01653509
Title: An Exploratory Study to Investigate the Inflammatory Response During a Cold Sore Episode
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Labtec GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E7411153
Record Dates: First submitted 2012-07-19; First posted 2012-07-31 (Estimated); Results first posted 2014-03-10 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-02

CONDITIONS: Herpes Labialis
Keywords: cold sore
MeSH Terms: conditions — Herpes Labialis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test patch (Experimental): Patch containing acyclovir applied to cold sore
  Interventions: Device: Acyclovir patch
- Placebo patch (Placebo Comparator): Patch without acyclovir applied to cold sore
  Interventions: Device: Placebo patch

INTERVENTIONS:
Device: Acyclovir patch — Patch containing acyclovir
  Arms: Test patch
Device: Placebo patch — Patch without acyclovir
  Arms: Placebo patch

SUMMARY:
This study will treat approximately 24 participants who experience cold sores. Patches will be applied to the cold sore for up to ten days, and the symptoms will be measured during daily clinic visits using non-invasive measurement techniques.

ELIGIBILITY:
Participants who are susceptible to cold sores that reactivate when exposed to ultraviolet (UV) light

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- proDERM Institute for Applied Dermatological Research GmbH, Hamburg, Germany

REFERENCES:
- [Derived] Veltri J, Boon R, Bohling A, Wilhelm KP, Bielfeldt S. A Randomized Exploratory Study to Investigate the Inflammatory Response During an Ultraviolet-Radiation-Induced Cold Sore Episode. Dermatol Ther (Heidelb). 2021 Jun;11(3):983-994. doi: 10.1007/s13555-021-00531-x. Epub 2021 Apr 28. PMID 33913104

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: 105 screened, 60 underwent ultraviolet (UV) rays induction, 25 developed a cold sore and were randomized into the study.
Groups:
- Acyclovir Patch: Participants applied single patch containing acyclovir to the cold sore area. A maximum of 5 patches/ day were allowed during the 10 day study period.
- Placebo Patch: Participants applied single placebo patch to the cold sore area. A maximum of 5 patches/ day were allowed during the 10 day study period.
Period: Overall Study
Arm/Group | Acyclovir Patch | Placebo Patch
Started | 12 | 13
Completed | 12 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Acyclovir Patch: Participants applied single patch containing acyclovir to the cold sore area. A maximum of 5 patches/ day were allowed during the 10 day study period. Baseline measures were determined for Safety population.
- Placebo Patch: Participants applied single placebo patch to the cold sore area. A maximum of 5 patches/ day were allowed during the 10 day study period. Baseline measures were determined for Safety population.
- Total: Total of all reporting groups
Arm/Group | Acyclovir Patch | Placebo Patch | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.6 (14.88) | 43.2 (15.60) | 45.3 (15.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Blood Flow
Description: Measurement of blood flow was performed using Field Laser Perfusion Imaging (FLPI) technique.
  Total episode value (TEV) was calculated as the summation of (test region response minus control region response) across all days. Maximum episode value (MEV) was calculated as the maximum of (test region response minus control region response) across all days.
Time Frame: Baseline to Day 10
Population: Intent to Treat (ITT) population: all randomized participants who had a patch applied to their cold sore and have at least one post-baseline efficacy measurement.
Measure: Least Squares Mean (Standard Error); unit: Perfusion Units
Arm/Group | Acyclovir Patch | Placebo Patch
Number analyzed (Participants) | 12 | 13
Perfusion Units
  TEV (Day 1 to Day 10) | 2558.65 (627.87) | 3470.13 (603.23)
  MEV | 809.88 (127.93) | 960.86 (122.91)
Statistical Analysis 1: Comparison: Acyclovir Patch vs Placebo Patch; Null hypothesis considered no difference between study treatments for TEV; Test type: Superiority or Other; p = 0.3061, ANOVA; ANOVA model with a factor for treatment group; Least square mean difference = -911.48, 95% CI 2-sided [-2712.65 to 889.69] — Difference calculated as first named treatment minus second named treatment, such that a negative difference favours the first named treatment
Statistical Analysis 2: Comparison: Acyclovir Patch vs Placebo Patch; Null hypothesis considered no difference between treatments for MEV; Test type: Superiority or Other; p = 0.4035, ANOVA; ANOVA model with a factor for treatment group; LS Mean Difference = -150.99, 95% CI 2-sided [-517.97 to 215.99] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Mean Change From Baseline in Temperature
Description: Lesion thermographic parameters for TEV and MEV were analysed.
Time Frame: Baseline to Day 10
Population: ITT population: all randomized participants who had a patch applied to their cold sore and have at least one post-baseline efficacy measurement.
Measure: Least Squares Mean (Standard Error); unit: Degree celsius
Arm/Group | Acyclovir Patch | Placebo Patch
Number analyzed (Participants) | 12 | 13
Degree celsius
  TEV (Day 1 to Day 10) | 3.24 (0.86) | 0.76 (0.82)
  MEV | 0.90 (0.15) | 0.51 (0.15)
Statistical Analysis 1: Comparison: Acyclovir Patch vs Placebo Patch; Null hypothesis considered no difference between study treatments for TEV (Day 1 to day 10); Test type: Superiority or Other; p = 0.0486, ANOVA; ANOVA model with a factor for treatment group; LS Mean Difference = 2.48, 95% CI 2-sided [0.02 to 4.93] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Acyclovir Patch vs Placebo Patch; Null hypothesis considered no difference between study treatments for MEV; Test type: Superiority or Other; p = 0.0799, ANOVA; ANOVA model with a factor for treatment group; LS Mean Difference = 0.38, 95% CI 2-sided [-0.05 to 0.82] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Mean Change From Baseline in Color Intensity of Lesions
Description: The redness of the cold sores to be measured and quantified using sophisticated, standardized and reproducible color photography. Parameter represents distance between test and control values according to a* axis and b* axis colour intensity values. The values on the scale ranged from -100 (green, lowest intensity) to +100 (red, highest intensity).
Time Frame: Baseline to Day 10
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Acyclovir Patch | Placebo Patch
Number analyzed (Participants) | 12 | 13
Units on a scale
  TEV | 11.05 (1.12) | 8.91 (1.07)
  MEV | 2.66 (0.22) | 2.29 (0.21)
Statistical Analysis 1: Comparison: Acyclovir Patch vs Placebo Patch; Null hypothesis considered no difference between study treatments for TEV; Test type: Superiority or Other; p = 0.1790, ANOVA; ANOVA model with a factor for treatment group; LS mean difference = 2.14, 95% CI 2-sided [-1.06 to 5.35] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Acyclovir Patch vs Placebo Patch; Null hypothesis considered no difference between study treatments for MEV; Test type: Superiority or Other; p = 0.2446, ANOVA; ANOVA model with a factor for treatment group; LS mean difference = 0.37, 95% CI 2-sided [-0.27 to 1.00] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Participant Assessment of Patch Comfort and Noticeability at Day 5
Description: Participants reported experience of the patch aesthetics and cold sore noticeability on the cold sore using a 5-point scale ( 1=Strongly Disagree 2=Rather Disagree 3=Neither Agree nor Disagree 4=Mostly Agree 5=Completely Agree) on 9 questions asked to them:
  1. Today my sore felt completely protected
  2. Today my cold sores interfered with facial movements such as smiling, eating or drinking
  3. Today my cold sores interfered with my interaction with other people
  4. Today the patch disguised my cold sores
  5. Today I was bothered by the appearance of my cold sores
  6. Today my patch was easy to apply
  7. Today the patch covering my cold sores was bothersome
  8. Today the patches stayed in place on my cold sores until I removed them
  9. Today the patches were easy to remove from my lip or skin
Time Frame: Day 5
Population: ITT population: all randomized participants who had a patch applied to their cold sore and had at least one post-baseline efficacy measurement. There were difference in number of participants analyzed for each end point as represented by "n".
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Acyclovir Patch | Placebo Patch
Number analyzed (Participants) | 12 | 13
Units on a scale
  Protection (n = 11, 12) | 4.45 (0.69) | 4.17 (1.12)
  Facial Movements (n = 11, 12) | 2.18 (1.33) | 2.75 (1.60)
  Interpersonal Interaction (n = 11, 12) | 2.09 (1.45) | 1.75 (0.97)
  Cold Sore Cover (n = 11, 12) | 4.45 (0.93) | 3.92 (1.31)
  Cold sore appearance (n = 11, 12) | 1.55 (0.93) | 1.67 (1.16)
  Ease of application (n = 11, 12) | 4.55 (0.69) | 4.00 (1.04)
  Bothersomeness (n = 11, 12) | 1.55 (0.93) | 1.55 (0.45)
  Adhesivenes (n = 11, 12) | 4.36 (0.92) | 3.75 (0.97)
  Patch removal (n = 9, 10) | 4.33 (1.00) | 4.60 (0.52)

5. Secondary Outcome: Participant Assessment of Patch Comfort and Noticeability at Day 10
Description: as for outcome 4
Time Frame: Day 10
Population: ITT population: all randomized participants who had a patch applied to their cold sore and have at least one post-baseline efficacy measurement. There were differences in number of participants analyzed for each end point as represented by "n".
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Acyclovir Patch | Placebo Patch
Number analyzed (Participants) | 12 | 13
Units on a scale
  Protection (n= 4, 7) | 4.50 (1.00) | 4.14 (1.07)
  Facial Movements (n= 4, 7) | 1.50 (1.00) | 2.29 (1.11)
  Interpersonal Interaction (n= 4, 7) | 1.50 (0.58) | 1.14 (0.38)
  Cold Sore Coverage (n= 4, 7) | 4.75 (0.50) | 4.57 (0.54)
  Cold sore appearance (n= 4, 7) | 1.50 (0.58) | 1.14 (0.38)
  Ease of application (n= 4, 7) | 4.75 (0.50) | 4.86 (0.38)
  Bothersomeness (n= 4, 7) | 1.50 (1.00) | 2.43 (1.40)
  Adhesiveness (n= 4, 7) | 4.75 (0.50) | 3.86 (1.35)
  Patch removal (n = 3, 5) | 4.33 (0.58) | 4.60 (0.89)

6. Secondary Outcome: Participant Assessment of Symptom Intensity at Day 5
Description: Cold sore symptoms (pain, burning, itching) assessment was evaluated on a 5-point scale: 1=Never Bothered, 2=Rarely Bothered, 3=Bothered Some of the Time, 4=Bothered Often, 5=Bothered All the Time.
Time Frame: Day 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Acyclovir Patch | Placebo Patch
Number analyzed (Participants) | 12 | 13
Units on a scale
  Pain/Soreness (n = 11, 12) | 1.55 (0.82) | 1.75 (1.22)
  Itching (n = 11, 12) | 1.18 (0.41) | 1.67 (0.99)
  Burning (n = 11, 12) | 1.36 (0.67) | 1.42 (0.67)

7. Secondary Outcome: Participant Assessment of Symptom Intensity at Day 10
Description: Cold sore symptoms (pain, burning, itching) assessment was performed on a 5-point scale: 1=Never Bothered 2=Rarely Bothered 3=Bothered Some of the Time 4=Bothered Often 5=Bothered All the Time.
Time Frame: Day 10
Population: ITT population: all randomized participants who had a patch applied to their cold sore and have at least one post-baseline efficacy measurement. There were differences in the number of participants analyzed for each end point, as represented by "n".
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Acyclovir Patch: Participants applied single patch containing acyclovir to the cold sore area at a time. A maximum of 5 patches/ day were allowed during the 10 day study period.
- Placebo Patch: Participants applied single placebo patch to the cold sore area at a time. A maximum of 5 patches/ day were allowed during the 10 day study period.
Arm/Group | Acyclovir Patch | Placebo Patch
Number analyzed (Participants) | 12 | 13
Units on a scale
  Pain/Soreness (n = 4, 7) | 1.00 (0.00) | 1.29 (0.49)
  Itching (n = 4, 7) | 1.00 (0.00) | 1.14 (0.38)
  Burning (n = 4, 7) | 1.00 (0.00) | 1.00 (0.00)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from UV exposure until the study completion assessments or the telephone follow-up for those participants not undergoing study completion assessments.
Groups:
- Acyclovir Patch: Participants applied single patch containing acyclovir to the cold sore area.
- Placebo Patch: Participants applied single placebo patch to the cold sore area.
Arm/Group | Acyclovir Patch | Placebo Patch
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 3/13
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acyclovir Patch (N=12) | Placebo Patch (N=13)
Lip Erosion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral Herpes (Infections and infestations) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was not formally powered to detect statistically significant differences, but to provide information for methods development and develop sample size calculation for future studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.